CLINICAL TRIAL: NCT00703482
Title: A Randomised, Double-Blind, Placebo-Controlled Study Assessing the Effect of Fenofibrate, Coenzyme Q10 and Their co-Administration on Ventricular Diastolic Function in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Solvay Pharmaceuticals (Industry)
Responsible Party: Jean Claude Ansquer, Solvay Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CFEN0205
Record Dates: First submitted 2008-06-20; First posted 2008-06-23 (Estimated); Last update posted 2008-06-25 (Estimated); Status verified 2008-06

CONDITIONS: Patients With Type 2 Diabetes
Keywords: Ventricular diastolic Function; Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Fenofibrate; coenzyme Q10

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (7):
- 1 (Placebo Comparator)
  Interventions: Drug: Fenofibrate/CoQ10
- 2 (Active Comparator)
  Interventions: Drug: Fenofibrate/CoQ10
- 3 (Active Comparator)
  Interventions: Drug: Fenofibrate/CoQ10
- 4 (Experimental)
  Interventions: Drug: Fenofibrate/CoQ10
- 5 (Experimental)
  Interventions: Drug: Fenofibrate/CoQ10
- 6 (Experimental)
  Interventions: Drug: Fenofibrate/CoQ10
- 7 (Experimental)
  Interventions: Drug: Fenofibrate/CoQ10

INTERVENTIONS:
Drug: Fenofibrate/CoQ10 — Fenofibrate pbo/CoQ10 placebo
  Arms: 1
Drug: Fenofibrate/CoQ10 — Fenofibrate pbo/CoQ10 200 mg
  Arms: 2
Drug: Fenofibrate/CoQ10 — Fenofibrate 160mg/CoQ10 placebo
  Arms: 1; 3
Drug: Fenofibrate/CoQ10 — Fenofibrate 80/CoQ10 100 mg
  Arms: 4
Drug: Fenofibrate/CoQ10 — Fenofibrate 160mg/CoQ10 100 mg
  Arms: 5
Drug: Fenofibrate/CoQ10 — Fenofibrate 80 /CoQ10 200 mg
  Arms: 6
Drug: Fenofibrate/CoQ10 — Fenofibrate 160mg/CoQ10 200 mg
  Arms: 7

SUMMARY:
The purpose of this study was to study the effect of different combinations of fenofibrate and coenzyme Q10 on ventricular diastolic function in patients with Type II diabetes

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged from 40 to 79 years
* Patients with pre-existing T2DM
* HbA1C <9%
* Written informed consent

Exclusion Criteria:

* unable to comply with the protocol, Likely to leave the trial before completion
* having participated in an another trial 3à days before V1
* Pregnant or childbearing potential not using birth control method
* Type 1 diabetic patients, T2Dm insulin therapy

Patients with one of the following pathology:

* with muscular disorders known or increase CK , or hepatic deficiency or transaminase increase
* with symptomatic gall-bladder disease or/and renal insufficiency
* with abnormal thyroid function
* with proliferative retinopathy
* with recent cardiovascular event, uncontrolled hypertension
* with known chronic alcohol intake
* with other severe pathology
* with TC>= 7.0 mmol/L and/or TG>= 4mmol/L at V1
* Patients treated with Warfarin
* Patients with specific ECG dysfunction

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2003-05; Primary Completion 2004-09 (Actual); Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Evolution of the E'/E septal ratio | End of study (V6)

SECONDARY OUTCOMES:
Severity of the LVDD | End of study (V6)
Evolution of the Left atrium and right atrium volumes | End of study (V6)
Evolution of the Left and right sizes | End of study (V6)
Evolution of the LVEDD and LVESD | End of study (V6)
Evolution of the LVEDV and LVESV | End of study (V6)
Evolution of the LV mass | End of study (V6)
Evolution of the LV ejection fraction | End of study (V6)
Evolution of the IVRT | End of study (V6)
Evolution of the tissue Doppler E'/A' ratio | End of study (V6)
Evolution of the PV doppler parameters | End of study (V6)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (3):
- Australia (3):
  - Site 002, Fremantle
  - Site 003, Nedlands
  - Site 001, Perth